CLINICAL TRIAL: NCT03996200
Title: A Prospective, Open, Multicentre Clinical Trial Analysing the Efficacy and Safety of Miniject (MINI SO627) in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications Using a Single Operator Delivery Tool
Brief Title: MINIject in Patients With Open Angle Glaucoma Using Single Operator Delivery Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-III (ISM08)
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma, Open-Angle; Glaucoma Eye
Keywords: glaucoma; medical device; MIGS; drainage device; eye; reduction IOP
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Intervention Model Description: MINIject SO627
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MINIject CS627 implant (Experimental): MINIject 627 implant is used to reduce intra-ocular pressure in the eye. It is implanted through a minimally-invasive glaucoma surgical intervention in a stand alone procedure.
  Interventions: Device: MINIject CS627 implant

INTERVENTIONS:
Device: MINIject CS627 implant — MINI SO627 is an integrated system comprising a minimally-invasive Glaucoma Drainage Implant (CS627) and a single operator delivery tool.
  The delivery tool is a single-use tool, designed for inserting the CS627 implant into the suprachoroidal space in the eye.

SUMMARY:
Study to assess safety and performance of MINIject SO627 in patients with open angle glaucoma.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of MINI SO627 and IOP (Intra- ocular pressure) lowering effects with or without the use of glaucoma medications. The procedure will be a stand alone surgery. Patient follow up with several examinations up to 24 months after surgery.

The primary endpoint is the reduction in medicated mean diurnal IOP at 6 months follow up compared to medicated diurnal IOP at baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary open angle glaucoma during screening/baseline visit or earlier.
* Grade 3 or grade 4 according to Shaffer Angle Grading System.
* Glaucoma not adequately controlled by one to four different topical hypotensive medication(s), given each for at least one month, as confirmed by 21mmHg < IOP < 35 mmHg in the study eye at baseline visit.

Exclusion Criteria:

* Grade 2 (narrow, 20 degrees), grade 1 (extremely narrow, less or equal to 10 degrees) and grade 0 (closed or slit) according to Shaffer Angle Grading System in the study eye.
* Neovascular glaucoma in the study eye.
* Corneal opacity or iridocorneal angle not visible through gonioprism in the study eye, preventing correct placement of the implant in the stud eye.
* Prior glaucoma surgery in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
medicated diurnal IOP | 6 months post surgery
  Change in medicated diurnal IOP

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR
Locations (3):
- Clinica Oftalmologica del Caribe, Barranquilla, Colombia
- Maxivision Eye Hospital, Hyderabad, Telangana, India
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No